CLINICAL TRIAL: NCT03629652
Title: Head-dOwn Position for ischEmic Stroke With Middle Cerebral Artery (HOPES): a Prospective, Random, Multi-Center, Pilot Trial
Brief Title: Head-dOwn Position for ischEmic Stroke With Middle Cerebral Artery (HOPES)
Acronym: HOPES
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: it is hard to enroll the patients
Sponsor: General Hospital of Shenyang Military Region (Other)
Responsible Party: Principal Investigator, Hui-Sheng Chen, Director of neurological department, General Hospital of Shenyang Military Region
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: k(2018)25
Record Dates: First submitted 2018-08-06; First posted 2018-08-14 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Ischemic Stroke
Keywords: head-down position; ischemic stroke; rehabilitation
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Head down position (Experimental): head-down position treatment combined with conventional rehabilitation.
  Interventions: Other: head-down position treatment; Other: Conventional Rehabilitation
- Conventional Rehabilitation (Sham Comparator): Conventional rehabilitation treatment
  Interventions: Other: Conventional Rehabilitation

INTERVENTIONS:
Other: head-down position treatment — In the head-down position, the body is in the supine position with the head lowered to 30 degrees
  Arms: Head down position
Other: Conventional Rehabilitation — The body is in the supine position without lowered head

SUMMARY:
The study is designed to explore the efficacy and safety of head-down position in patients with acute ischemic stroke。

DETAILED DESCRIPTION:
Currently, the guideline recommended re-perfusion such as intravenous thrombolysis and mechanical thrombectomy as the most effective treatment for acute ischemic stroke. However, the two methods are restricted by a strict time window, which greatly limits the number of the patients receiving treatment. The abundant studies have suggested that good collateral circulation can provide compensatory blood supply to save the ischemic penumbra and reduces the infarct volume, which improves the prognosis. How to improve collateral circulation in an efficient and safe way is a clinical challenge. Our recent experiment results of the animal and clinical experiments show that head-down position can significantly increase cerebral perfusion and improve neurological function. Clinically, head-down position is simple and easy to operate, and theoretically may increases brain perfusion and improve collateral circulation. A pilot randomized clinical trial is designed to investigate the effect of head-down position combined with routine rehabilitation in patients with ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥18 years
2. acute ischemic stroke within 10 - 30 days of onset
3. neurological deficit: 6≤NIHSS≤16
4. Large artery atherosclerosis stroke based on TOAST criteria
5. The responsibility vessels were the middle cerebral artery or internal carotid artery, and the degree of stenosis was more than 50%.
6. first stroke onset or past stroke without obvious neurological deficit (mRS≤1)
7. fully understand and cooperate with the doctor's instructions.
8. the availability of informed consent;

Exclusion Criteria:

1. Hemorrhagic stroke or mixed stroke
2. Combining with severe organ dysfunction
3. Past hemorrhagic stroke
4. A history of stroke with severe sequelae
5. Planning revascularization in 3 months
6. Ischemic stroke due to surgical intervention
7. participating in other clinical trials within 3 months
8. Pregnant or lactating women
9. any inappropriate patients assessed by the researcher

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-08-06 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
proportion of patients with modified Rankin Score 0 to 2 | 90 days

SECONDARY OUTCOMES:
proportion of patients with modified Rankin Score 0 to 1 | 90 days
The percentage of reduction in Fugl-Meyer score | 90 days
occurrence of stroke | 90 days
  stroke or TIA
The percentage of reduction in MMSE | 90 days
  MMSE，Mini-mental State Examination
The percentage of reduction in MoCA | 90 days
  MoCA, Montreal Congnitive Assessment
Incidence of major vascular events | 90 days
  ischemic stroke, hemorrhagic stroke, TIA, myocardial infarction, vascular death
the biggest tolerance time of head-down | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Sheng Chen, doctor, Principal Investigator — General Hospital of Shenyang Military Region
Locations (1):
- General Hospital of ShenYang Military Region, Shenyang, Liaoning, China